CLINICAL TRIAL: NCT07186374
Title: Relationship of Radiographic Findings With Pain, Function, Physical Performance and Balance in Patients With Hip Osteoarthritis
Brief Title: Relationship of Radiographic Findings With Pain, Function, Physical Performance and Balance
Status: Recruiting | Type: Observational
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Zeynep Yıldız Kızkın, Lecturer, Artvin Coruh University
Other Study IDs: Hip Osteoarthritis
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Hip Osteoarthritis
Keywords: hip; osteoarthritis; function; balance; radiography
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Hip Osteoarthritis (PwHOA): Adults diagnosed with hip osteoarthritis will be included in the study.

SUMMARY:
The objective of this investigation was to examine the correlation between radiographic findings and clinical outcomes, including pain, functional ability, physical performance, and balance parameters, in patients diagnosed with hip osteoarthritis (PwHOA).

DETAILED DESCRIPTION:
A total of seventy-two patients with hip osteoarthritis (PwHOA) will be enrolled in the study. Sociodemographic variables will be collected, and assessments will include the Kellgren-Lawrence Classification, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Timed Up and Go Test (TUG), and Four Square Step Test (FSST). The Spearman rank correlation coefficient will be employed to analyze the relationships among pain levels, functional capacity, physical performance, balance, and radiographic findings.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic and radiographic diagnosis of Grade I-IV hip osteoarthritis according to the Kellgren-Lawrence classification and American College of Rheumatology criteria.

Exclusion Criteria:

* patients who did not give consent to participate in the study;
* secondary HOA due to rheumatoid arthritis, tumors, and recent fractures;
* history of intra-articular injections within the last six months.

Ages: 40 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with hip osteoarthritis will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Kellgren-Lawrence Classification | Single assessment at enrollment
  This assessment, acknowledged by the World Health Organization as the definitive standard for the radiographic classification of osteoarthritis, shall be conducted by a qualified orthopaedic specialist. The evaluation will be based on radiographic imaging obtained in both the sagittal and frontal planes while the patient maintains an upright stance. Utilizing the 0-4 severity grading system, a score of '0' denotes the absence of osteoarthritis, whereas a score of '4' signifies advanced, severe osteoarthritic changes.
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Single assessment at enrollment
  This index, employed for the evaluation of pain, stiffness, and functional impairment, has demonstrated validity and reliability in patients diagnosed with Knee Osteoarthritis (KOA) and Hip Osteoarthritis (HOA), with Intraclass Correlation Coefficients (ICC) ranging from 0.80 to 0.90. It comprises 24 items, each rated on a 5-point Likert scale from 0 to 4, where 0 indicates absence of symptoms, 1 signifies mild symptoms, 2 denotes moderate severity, 3 corresponds to severe symptoms, and 4 reflects extreme severity.
Timed Up and Go Test (TUG) | Single assessment at enrollment
  The procedure will initiate with participants seated upright in a chair with their arms resting on their laps. The time required for each participant to rise from a chair elevated to 45 centimeters, traverse a distance of 3 meters at maximum effort, execute a turnaround, and return to the original chair to sit will be measured in seconds utilizing a stopwatch. Following a preliminary trial, the mean duration from two recorded trials will be calculated for analysis.
Four Square Step Test | Single assessment at enrollment
  The assessment of dynamic balance will be conducted utilizing the four-square step test. The test environment will be delineated by arranging bars, each measuring 90 cm in length, in a '+' configuration. The squares will be sequentially numbered clockwise from 1 to 4, commencing with the bottom left square. Participants will be instructed to traverse the squares following the sequence: 2 → 3 → 4 → 1 → 4 → 3 → 2 → 1. The time required to complete the sequence will be measured in seconds using a stopwatch. Following an initial practice trial, the average of two recorded trials will be calculated for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Yıldız Kızkın, Dr., Principal Investigator — Artvin Coruh University
Locations (1):
- Zeynep Yıldız Kızkın, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson AE, Hu D, Arbeeva L, Alvarez C, Cleveland RJ, Schwartz TA, Murphy LB, Helmick CG, Callahan LF, Renner JB, Jordan JM, Golightly YM. Point prevalence of Hip Symptoms, Radiographic, And Symptomatic OA at Five Time Points: The Johnston County Osteoarthritis Project, 1991-2018. Osteoarthr Cartil Open. 2022 Jun;4(2):100251. doi: 10.1016/j.ocarto.2022.100251. Epub 2022 Mar 15. PMID 36118130
- [Background] Turkiewicz A, Kiadaliri AA, Englund M. Cause-specific mortality in osteoarthritis of peripheral joints. Osteoarthritis Cartilage. 2019 Jun;27(6):848-854. doi: 10.1016/j.joca.2019.02.793. Epub 2019 Feb 21. PMID 30797945
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Background] Ritsuno Y, Morita M, Mukaino M, Otsuka K, Kanaji A, Yamada J, Saitoh E, Matsumoto M, Nakamura M, Otaka Y, Fujita N. Determinants of Gait Parameters in Patients With Severe Hip Osteoarthritis. Arch Phys Med Rehabil. 2024 Feb;105(2):343-351. doi: 10.1016/j.apmr.2023.08.021. Epub 2023 Sep 7. PMID 37683907
- [Background] Ozden F, Nadiye Karaman O, Tugay N, Yalin Kilinc C, Mihriban Kilinc R, Umut Tugay B. The relationship of radiographic findings with pain, function, and quality of life in patients with knee osteoarthritis. J Clin Orthop Trauma. 2020 Jul;11(Suppl 4):S512-S517. doi: 10.1016/j.jcot.2020.04.006. Epub 2020 Apr 9. PMID 32774020
- [Background] Jacobsen S. Adult hip dysplasia and osteoarthritis. Studies in radiology and clinical epidemiology. Acta Orthop Suppl. 2006 Dec;77(324):1-37. PMID 17380595
- [Background] Riddle DL, Perera RA. American Academy of Orthopedic Surgeons Appropriate Use Criteria for Hip Preservation Surgery: Variables That Drive Appropriateness for Surgery. Arthritis Care Res (Hoboken). 2020 Mar;72(3):405-411. doi: 10.1002/acr.23828. PMID 30675763
- [Background] Hattori T, Shimo K, Niwa Y, Tokiwa Y, Matsubara T. Association of Chronic Pain with Radiologic Severity and Central Sensitization in Hip Osteoarthritis Patients. J Pain Res. 2021 Apr 22;14:1153-1160. doi: 10.2147/JPR.S296273. eCollection 2021. PMID 33911897
- [Background] Rondas GA, Macri EM, Oei EH, Bierma-Zeinstra SM, Rijkels-Otters HB, Runhaar J. Association between hip pain and radiographic hip osteoarthritis in primary care: the CHECK cohort. Br J Gen Pract. 2022 Jul 26;72(723):e722-8. doi: 10.3399/BJGP.2021.0547. Online ahead of print. PMID 36127152
- [Background] Pereira D, Severo M, Santos RA, Barros H, Branco J, Lucas R, Costa L, Ramos E. Knee and hip radiographic osteoarthritis features: differences on pain, function and quality of life. Clin Rheumatol. 2016 Jun;35(6):1555-64. doi: 10.1007/s10067-015-3087-7. Epub 2015 Oct 7. PMID 26445941
- [Background] Cubukcu D, Sarsan A, Alkan H. Relationships between Pain, Function and Radiographic Findings in Osteoarthritis of the Knee: A Cross-Sectional Study. Arthritis. 2012;2012:984060. doi: 10.1155/2012/984060. Epub 2012 Nov 19. PMID 23209900
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Iidaka T, Horii C, Muraki S, Oka H, Kawaguchi H, Nakamura K, Akune T, Tanaka S, Yoshimura N. Trends in prevalence of hip osteoarthritis over a 10-year period in Japan: The ROAD study 2005-2015. Osteoarthr Cartil Open. 2022 Jun 22;4(3):100285. doi: 10.1016/j.ocarto.2022.100285. eCollection 2022 Sep. PMID 36474937
- [Background] Batting M, Barker KL. Reliability and validity of the Four Square Step Test in patients with hip osteoarthritis before and after total hip replacement. Physiotherapy. 2019 Jun;105(2):244-253. doi: 10.1016/j.physio.2018.07.014. Epub 2018 Oct 15. PMID 30630621
- [Background] Canzone A, Roggio F, Patti A, Giustino V, Mannucci C, Di Mauro D, Musumeci G, Bianco A, Trimarchi F. Classification of Physical Activity Programs Based on the Kellgren & Lawrence Scale for Knee Osteoarthritis: A Systematic Review. Musculoskeletal Care. 2024 Dec;22(4):e70019. doi: 10.1002/msc.70019. PMID 39592397
- [Background] Thumboo J, Chew LH, Soh CH. Validation of the Western Ontario and Mcmaster University osteoarthritis index in Asians with osteoarthritis in Singapore. Osteoarthritis Cartilage. 2001 Jul;9(5):440-6. doi: 10.1053/joca.2000.0410. PMID 11467892
- [Background] Alghadir A, Anwer S. Effect of retro and forward walking on quadriceps muscle strength, pain, function, and mobility in patients with knee osteoarthritis: a protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2016 Apr 12;17:161. doi: 10.1186/s12891-016-1021-z. PMID 27072798